CLINICAL TRIAL: NCT05180357
Title: Retrospective, Observational Study in Patients With Severe Eosinophilic Asthma and Nasal Polyps Treated by FASENRA®
Brief Title: RANS. Study in Patients With Severe Eosinophilic Asthma and Nasal Polyps.
Acronym: RANS
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D3250R00099
Record Dates: First submitted 2021-10-14; First posted 2022-01-06 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Severe Eosinophilic Asthma; Nasal Polyps
Keywords: Severe Eosinophilic Asthma, nasal polyps, benralizumab, FASENRA.
MeSH Terms: conditions — Pulmonary Eosinophilia; Nasal Polyps | interventions — benralizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- SEA+NP Patients on FASENRA (benralizumab): SEA+NP Patients on FASENRA (benralizumab)
  Interventions: Other: FASENRA(benralizumab)

INTERVENTIONS:
Other: FASENRA(benralizumab) — This is a retrospective, observational study with secondary data collection utilizing medical chart review in hospitals or clinical centres that treated SEA + NP patients with benralizumab. Patient data including demographics, clinical characteristics, medication history, biologic treatment, and NP and asthma clinical outcomes will be abstracted from patient medical charts onto a pre-approved electronic case report form. No personal identifiable data will be collected. Data from all participating centres will be combined into a single anonymised dataset for analysis.

SUMMARY:
The purpose of this observational study is to describe the population of patients with SEA + NP who have been prescribed FASENRA and assess available clinical outcomes for both NP and asthma.

DETAILED DESCRIPTION:
In light of the increasing importance of comorbidities in driving choice for biologics in severe asthma there is a knowledge gap to understand SEA patients with comorbid NP for whom the decision to start biologics was based on the presence of severe, uncontrolled asthma. This retrospective, observational study will describe the population of patients with SEA + NP who have been prescribed FASENRA and assess available clinical outcomes for both NP and asthma.

ELIGIBILITY:
Inclusion Criteria:

1. Current or previous treatment with benralizumab for SEA
2. Physician-confirmed diagnosis and evaluation of NP using NPS and/or SNOT-22 before and after first benralizumab injection
3. Patients who have follow-up period of at least 5 months from first benralizumab injection or at least 4 consecutive injections of benralizumab
4. Able to provide signed informed consent (if required based on local guidelines)

Exclusion Criteria:

1. Patient on any other biologic during the 12 months prior to treatment with benralizumab
2. Previously or currently receiving any biologics for the treatment of asthma or NP in a clinical trial. This exclusion criteria does not apply to patients that received biologic treatment from openlabel one-arm interventional studies that provided biologic treatment as part of standard of care (according to approved labelling in that country).

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is SEA + NP patients on benralizumab.
Sampling Method: Non-Probability Sample
Enrollment: 273 (Actual)
Dates: Start 2021-11-23 (Actual); Primary Completion 2022-10-28 (Actual); Study Completion 2022-10-28 (Actual)

PRIMARY OUTCOMES:
Baseline demographics, clinical characteristics, and background treatments, as well as PROs for asthma control and HRQoL, asthma exacerbation, and healthcare resource utilization. | At or up to 12 months prior to first benralizumab dose.
  To describe baseline demographics, clinical characteristics, and background treatments, as well as PROs (patient-reported outcomes) for asthma control and HRQoL(health-related quality of life), asthma exacerbation, and healthcare resource utilization.

SECONDARY OUTCOMES:
Total NPS | Up to 12 months prior to and up to 12 months from first benralizumab dose.
  To describe the distribution (mean, median, range) of NPS (nasal polyp score) before and after initiation of benralizumab among SEA (severe eosinophilic asthma) +NP (nasal polyps) patient. NPS is the sum of the left and the right nostril scores evaluated by nasal endoscopy. Total score ranges from 0 to 8, with higher scores indicate larger-sized polyps.
SNOT-22 total score | Up to 12 months prior to and up to 12 months from first benralizumab dose.
  To describe the distribution (mean, median, range) of NP patient reported HRQoL total score (SNOT-22[Sino-nasal Outcome Test-22]) before and after initiation of benralizumab among EA+NP patients. SNOT-22 measures physical problems, functional limitations, and emotional consequences of sino-nasal conditions. SNOT-22 total score is calculated as the sum of all 22 responses and range from 0 to 110 (higher scores indicate poorer HRQoL).
Overall SCS use. SCS use for asthma only. SCS use for NP only | Up to 12 months from first benralizumab dose.
  To describe the use of SCS (systemic corticosteroids) after initiation of benralizumab among SEA + NP patients
Asthma Clinical outcomes. | Up to 12 months from first benralizumab dose.
  To describe asthma exacerbations, PROs, lung function, and benralizumab treatment patterns.
NP surgery type and/or procedure | Up to 12 months from first benralizumab dose.
  Proportion of patients with different type of surgery and/or procedure
Repeated or revision surgery for NP | Up to 12 months from first benralizumab dose.
  Proportion of patients with repeated or revision surgery
Time to NP surgery | Up to 12 months from first benralizumab dose.
  Timing (in days) from first benralizumab dose to NP surgery and/or repeated/revision surgery
NP surgery complications | Up to 12 months from first benralizumab dose.
  Proportion of patients with minor and major surgical complication.

OTHER OUTCOMES:
Asthma medications | Up to 12 months from first benralizumab dose.
  To describe asthma medications.
NP medications | Up to 12 months from first benralizumab dose.
  To describe NP medications.
All-cause healthcare resource utilization | Up to 12 months from first benralizumab dose.
  To describe all-cause healthcare resources utilization.
Asthma-related healthcare resources utilization | Up to 12 months from first benralizumab dose.
  To describe asthma-related healthcare resources utilization.
NPS by subgroups | Up to 12 months prior to and up to 12 months from first benzelizumab dose.
  To describe the distribution (mean, median) of NPS among subgroups of patients with different characteristics: demographics, clinical characteristics, and asthma clinical outcomes (number of exacerbations).
  NPS is the the sum of left and right nostril scores evaluated by nasal endoscopy. Total score ranges from 0 to 8, with higher scores indicate larger-sized polyps.
SNOT-22 total score by subgroups | Up to 12 months prior to and up to 12 months from first benralizumab dose.
  To describe the distribution (mean, median) of SNOT-22 total scores among subgroups of patients with different characteristics : demographics, clinical characteristics, and asthma clinical outcomes (number of exacerbations).
  SNOT-22 measures physical problems, functional limitations, and emotional consequences of sino-nasal conditions. SNOT-22 total score is calculated as the sum of all 22 responses and range from 0 to 110 (higher scores indicate poorer HRQoL).

CONTACTS AND LOCATIONS:
Locations (41):
- United States (8):
  - Research Site, Centennial, Colorado
  - Research Site, Denver, Colorado
  - Research Site, Glendale, New York
  - Research Site, New York, New York
  - Research Site, Rochester, New York
  - Research Site, The Bronx, New York
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Norfolk, Virginia
- France (5):
  - Research Site, Lyon
  - Research Site, Marseille
  - Research Site, Montpellier
  - Research Site, Nantes
  - Research Site, Strasbourg
- Germany (2):
  - Research Site, Lübeck
  - Research Site, Wiesbaden
- Italy (12):
  - Research Site, Catania
  - Research Site, Catanzaro
  - Research Site, Florence
  - Research Site, Milan
  - Research Site, Modena
  - Research Site, Monserrato
  - Research Site, Napoli
  - Research Site, Orbassano
  - Research Site, Ragusa
  - Research Site, Rome
  - Research Site, Salerno
  - Research Site, Varese
- Japan (6):
  - Research Site, Chuo-ku, Niigata-Shi
  - Research Site, Hiroshima
  - Research Site, Moriguchi-Shi
  - Research Site, Nagaoka-Shi
  - Research Site, Shinagawa-ku
  - Research Site, Yonago-Shi
- Spain (8):
  - Research Site, A Coruña
  - Research Site, Alcorcón
  - Research Site, Barcelona
  - Research Site, Cadiz
  - Research Site, Madrid
  - Research Site, Salamanca
  - Research Site, Seville
  - Research Site, Valencia

REFERENCES:
- [Derived] Le TT, Emmanuel B, Katial R, Tran TN, Kwiatek JJ, Cohen DS, Daniel SR, Cao Y, Shih VH, Melcon MG, Devouassoux G, Pelaia G; RANS Study Investigators. Benralizumab in Severe Eosinophilic Asthma and Chronic Rhinosinusitis with Nasal Polyps: The Real-World, Multi-Country RANS Observational Study. J Asthma Allergy. 2024 Apr 5;17:313-324. doi: 10.2147/JAA.S437190. eCollection 2024. PMID 38595692
- See also: CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D3250R00099&attachmentIdentifier=5be06e72-f9e5-4c8c-a6ba-c2db47af6bbe&fileName=d3250r00099-study-report-synopsis-redacted.pdf&versionIdentifier=